CLINICAL TRIAL: NCT01199211
Title: Impact of Physical Activity on Left Ventricular Mass and Lipid Metabolism in Healthy Female Volunteers Training for a Marathon
Brief Title: Impact of Physical Activity on Left Ventricular Mass and Lipid Metabolism
Status: Terminated | Type: Observational
Why Stopped: IRB approval expired
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: CTSI-6212
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2020-07-31 (Actual); Status verified 2020-07

CONDITIONS: Left Ventricular Hypertrophy
Keywords: hypertrophy, exercise, HDL, lipids, cholesterol
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Hypertrophy; Motor Activity | interventions — Exercise; Marathon Running

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Exercise training, women, marathon.: Other: prospective study with no intervention
  Interventions: Other: Exercise training, women, marathon

INTERVENTIONS:
Other: Exercise training, women, marathon — Prospective study with no intervention in women who have volunteered to run a full marathon or a half-marathon. Each subject will serve as own control. Each subject will be studies at 3 stages: baseline, after at least 12 weeks of training for the marathon (we will not provide training), 6 weeks after running the marathon.

SUMMARY:
Prospective study on the structural and functional changes in the heart of adult women assessed by echocardiogram and in lipid metabolism that occur in response to physical training. Using echocardiogram we will characterize the early determinants of "athletic remodeling". We will also assess the effect of intense physical training on lipid metabolism, focus on HDL subspecies and function.

DETAILED DESCRIPTION:
Left ventricular hypertrophy, defined as an increase in the mass of the left ventricle may occur as a physiologic response to exercise (athletic remodeling aka "athletic heart"), but is most frequently encountered as a pathological manifestation of cardiovascular disease. The early determinants of athletic remodeling in the general population are largely unknown. In order to longitudinally explore the early determinants of athletic remodeling, we will recruit from the community, physically untrained women who have volunteered to run a marathon. We will prospectively assess left ventricular mass and function by echocardiogram during three consecutive stages/visits:

* Baseline: prior to starting intense physical training
* Trained: at the end of at least 12 week training period, prior to running the marathon.
* Post-marathon: 6 weeks after running the marathon.

In addition, exercise impacts lipid metabolism and short-term exercise is known to increase HDL levels in plasma. Human HDL is structurally heterogeneous, comprising at least sixteen discrete species. It has multiple functions, pertinent to cardiovascular medicine such as the ability to accept effluxed cholesterol from the artery wall, culminating in sterol uptake in the liver. This "reverse cholesterol transport pathway" is thought to prevent the accumulation of cholesterol in the artery wall. We will assess the clinical and genetic determinants of the HDL response to physical exercise.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult men or women, aged 18 years or older
* Voluntarily signed up for a sport event or to run a marathon or a half marathon for the first time
* Normal to mildly elevated blood pressure (systolic blood pressure < 140 mmHg and/or diastolic blood pressure < 90 mmHg)
* Hormone replacement therapy and birth control pills are allowed, provided they have been on a stable dose for more than 3 months and no change in dose is planned for the duration of the study
* Capable and willing to provide written, informed consent for the study

Exclusion Criteria:

* History of cardiovascular disease within the past year (cardiomyopathy, heart failure, ischemic heart disease, stroke, TIA, peripheral vascular disease)
* Change in body weight more than 10% over the past year
* History of significant medical conditions, including respiratory, gastrointestinal, neuromuscular, neurological or musculoskeletal problems interfering with exercise.
* Autoimmune or collagen vascular diseases, chronic anemia,
* Malignancies in the past 5 years, with the exception of treated skin or breast cancer that did not require treatment with chemotherapy.
* Diabetes
* Pregnancy or recent delivery: delivery date less than 3 months prior to enrollment
* Lipid lowering medications (statins, niacin, resins) are allowed, provided dose has not changed for 3 months prior to enrollment and is not anticipated to change during the study
* Fish Oil supplements are allowed, provided dose has been unchanged for 3 months prior to enrollment and no change in dose is planned for the duration of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample. Participants will be recruited by invitation to volunteer in the study.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2011-02; Primary Completion 2017-10 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Lipid Metabolism | Baseline, In-Training, Post-training (at least 6 weeks after the race)

SECONDARY OUTCOMES:
Heart architecture and function | Baseline, In-training, Post-training

CONTACTS AND LOCATIONS:
Overall Officials: Eveline Stock, MD, Principal Investigator — University of California, San Francisco; Nelson Schiller, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- CTSI - University of California San Francisco, San Francisco, California, United States